CLINICAL TRIAL: NCT00599729
Title: Measurement of Gait Spatio-Temporal Characteristics in Knee Osteoarthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Prof. Nahum Halperin, Assaf-Harofeh Medical Center
Other Study IDs: 185/07; 185/07
Record Dates: First submitted 2008-01-14; First posted 2008-01-24 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2007-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patient demonstrating degenerative changes in the knee joint (osteoarthritis)

SUMMARY:
The purpose of the study is to evaluate the gait spatio-temporal parameters of patients with degenerative changes in the knee joint and to relate them with 2 questionares (WOMAC and SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee OA for at least 6 months
* Fulfilled American College of Rheumatology clinical criteria for OA of the knee
* Radiographically assessed OA of the knee graded 1-4 according to the Kellgren & Lawrence scale

Exclusion Criteria:

* Acute septic arthritis
* Patients with an increased tendency to fall
* Lack of physical or mental ability to perform or comply with the treatment procedure
* Diabetes mellitus
* History of pathological osteoporotic fracture

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with knee osteoarthritis evaluated by an orthopedic surgeon. patient will be recruted from the outpatient clinic at "asaf Harofe" medical center, Zrifin, Israel and APOS medical center, Herzlya, Israel
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nahum Halperin, Prof (MD), Study Chair — "asaf Harofe" Medical Center, Zrifin, Israel
Locations (2):
- Israel (2):
  - APOS Medical Center, Herzliya
  - "Asaf Harofeh" Medical center, Zrifin

REFERENCES:
- [Derived] Elbaz A, Mor A, Segal O, Agar G, Halperin N, Haim A, Debbi E, Segal G, Debi R. Can single limb support objectively assess the functional severity of knee osteoarthritis? Knee. 2012 Jan;19(1):32-5. doi: 10.1016/j.knee.2010.12.004. Epub 2011 Jan 26. PMID 21269835
- [Derived] Debi R, Mor A, Segal O, Segal G, Debbi E, Agar G, Halperin N, Haim A, Elbaz A. Differences in gait patterns, pain, function and quality of life between males and females with knee osteoarthritis: a clinical trial. BMC Musculoskelet Disord. 2009 Oct 13;10:127. doi: 10.1186/1471-2474-10-127. PMID 19825163